CLINICAL TRIAL: NCT01844128
Title: The Effect of Weight Loss on Ovarian Reserve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Amir Wiser, Senior physician IVF Unit, Meir Medical Center
Other Study IDs: 0257-12mmc
Record Dates: First submitted 2013-04-28; First posted 2013-05-01 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-04

CONDITIONS: Weight Loss
Keywords: MMA, AFC, Ovarian reserve
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- overweight women with infertility
  Interventions: Dietary Supplement: weight loss

INTERVENTIONS:
Dietary Supplement: weight loss

SUMMARY:
Obesity affects on fertility. Obese women have lower pregnancy rate after infertility treatments.They need more doses of hormone during ovarian stimulation, more days for stimulation. During IVF treatment less oocytes are collected and the quality of embryo also harmed.

The first line treatment for those women with obesity and infertility is weight loss.

The investigators' hypothesis is that weight reduction improves ovarian reserve and fertility treatment outcome.

DETAILED DESCRIPTION:
The investigators have outpatient clinic for obesity and infertility. the patients undergoing program of 3 months with diet and physical activity. Blood sample will take at the beginning of the program and at the end. The blood sample will evaluate for: AMH, Adiponectin, Leptin, CRP, Colesterol, CRP, Smac in addition TVUS will perform to evaluate AFC.

ELIGIBILITY:
Inclusion Criteria:

* undergoing weight loss program

Exclusion Criteria:

* dropp out before comletion the weighy loss target

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Overweight women with infertility
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Anti Mullerain Hormone (AMH)and AFC before and after weight loss | 3 months
  AMH and AFC will measure at the first visit and after 3 months of weight loss program

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel